CLINICAL TRIAL: NCT07330440
Title: A Phase I, Dose-escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of an mRNA Vaccine Against Herpes Simplex Virus Type 2 (HSV-2) in Healthy Participants Aged 18-55 Years, Stratified by Serostatus
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, and Immunogenicity of an mRNA Vaccine Against Herpes Simplex Virus Type 2 (HSV-2) Post-Vaccination
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B2101-F20240206-1
Record Dates: First submitted 2025-09-23; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Cohort Studies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo Group
- Low-Dose (Experimental): HSV-2 mRNA Vaccine
  Interventions: Biological: Low-Dose Cohort
- Mid-Dose (Experimental): HSV-2 mRNA Vaccine
  Interventions: Biological: Mid-Dose Cohort
- High-Dose (Experimental): HSV-2 mRNA Vaccine
  Interventions: Biological: High-Dose Cohort

INTERVENTIONS:
Biological: Low-Dose Cohort — Each human dose is 0.25 mL
  Arms: Low-Dose
Biological: Mid-Dose Cohort — Each human dose is 0.5 mL
  Arms: Mid-Dose
Biological: High-Dose Cohort — Each human dose is 1.0 mL
  Arms: High-Dose
Biological: Placebo Group — Each human dose: 0.25 mL, 0.5 mL, or 1.0 mL
  Arms: Placebo

SUMMARY:
A Preliminary Evaluation of the Safety and Immunogenicity Post-Vaccination with Different Doses of an mRNA Vaccine against Herpes Simplex Virus Type 2 (HSV-2) in Populations with Different Serostatus

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy male or female aged 18 to 55 years (inclusive) at the time of screening.
* Has provided written informed consent prior to performing any study-specific procedure.
* Is available and willing to comply with all study procedures for the entire duration of the study.
* For participants of childbearing potential: agrees to practice highly effective contraception for the required period and has no plans for reproduction or gamete donation.
* Provides consent for HSV-1/HSV-2 serology testing at screening.

Exclusion Criteria:

* Axillary temperature >37.0°C during screening and/or on the day of vaccination.
* History of clinically diagnosed genital herpes within 6 months prior to the first vaccination.
* Acute infectious disease or acute exacerbation of a chronic condition within 3 days prior to screening/vaccination.
* Positive blood pregnancy test at screening or currently breastfeeding (for female participants).
* History of severe allergic reactions requiring medical intervention (e.g., anaphylaxis, angioedema, Arthus reaction, allergic purpura), severe adverse reactions to previous vaccinations, or known hypersensitivity to any component of the investigational vaccine (e.g., lipid nanoparticles).
* Known or suspected malignancy, autoimmune disease, immunodeficiency, organ transplantation, or immunosuppression (e.g., HIV infection, systemic lupus erythematosus [SLE], rheumatoid arthritis).
* Use of immunosuppressants or immunomodulators (e.g., systemic corticosteroids for >14 consecutive days) or cytotoxic therapy within 6 months prior to the first vaccination, or planned use during the study.
* Congenital anomalies or developmental disorders affecting organ function.
* History of cardiovascular diseases (e.g., myocardial ischemia, myocardial infarction, myocarditis, pericarditis, idiopathic cardiomyopathy, arrhythmias), or any condition increasing the risk of myocarditis/pericarditis; QTcF >450 ms for males or >470 ms for females; or uncontrolled hypertension (systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg despite medication).
* For HSV-1/HSV-2 seronegative participants: clinically significant abnormalities in hematology, blood biochemistry, coagulation, or urinalysis parameters at screening.
* For HSV-1/HSV-2 seropositive participants: hematology, blood biochemistry, coagulation, or urinalysis parameters ≥ Grade 1 per the study-specific toxicity grading scale and deemed clinically significant by the investigator.
* Contraindications to intramuscular injection (e.g., thrombocytopenia, coagulation disorders).
* Medical conditions requiring intervention affecting the endocrine, hematologic, hepatic, renal, respiratory, metabolic, or skeletal systems.
* History of convulsions (excluding febrile seizures in childhood), epilepsy, encephalopathy, psychiatric disorders, or other neurological conditions; or family history of psychiatric disorders.
* Positive markers for HBV, HCV, HIV, or syphilis infection.
* Administration of blood products or immunoglobulins within 3 months prior to the first vaccination or planned use during the study.
* Treatment with anti-herpetic drugs (e.g., acyclovir, valacyclovir, famciclovir, ganciclovir) for genital herpes within 6 months prior to the first vaccination.
* Receipt of live-attenuated vaccines within 14 days, or subunit/inactivated vaccines within 7 days prior to vaccination.
* Participation in another clinical trial (drug, device, or vaccine) within 3 months prior to the first vaccination or concurrent enrollment in any interventional study.
* Any other condition deemed by the investigator to compromise participant safety or interfere with study objectives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-03-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoints | Up to 30 days after each dose
  Incidence of Adverse Events within 30 Days After Each Vaccination

SECONDARY OUTCOMES:
Safety Endpoints | from Day 0 up to 540 days
  The incidence of all Serious Adverse Events (SAEs)、Adverse Events of Special Interest (AESIs) from Day 0 until 12 months after the final vaccination
Safety Endpoints | up to 14 days
  Incidence of clinically significant abnormal electrocardiogram (ECG) findings after each vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Beijing, China